CLINICAL TRIAL: NCT03873740
Title: A Opened，Randomized and Controlled Trial to Evaluate the Immunity and Safety of Sequential Vaccination of Two Different Commercial EV71 Inactived Vaccines in Healthy Infants Aged 6-35 Months
Brief Title: Immunogenicity and Safety of Two Different Commercial EV71 Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Collaborators: Shandong Province Centers for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EV71-SD-2018-01
Record Dates: First submitted 2019-03-02; First posted 2019-03-13 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2019-03

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: Inactivated Enterovirus Type 71 (EV71) Vaccine; Sequential vaccination; Immunity; Safety
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single vaccine group A (Experimental): This group receive two doses injection of EV71 inactived vaccines(Vero cells) on Day 0 and 30, and two times of blood sampling on day of 0 and 60 respectively for EV71 neutralizing antibody detection.The vaccine was manufactured by Sinovac Vaccine Technology Co., Ltd.
  Interventions: Biological: EV71 inactived vaccine（Vero cells）
- Single vaccine group B (Experimental): This group receive two doses injection of EV71 inactived vaccines(human diploid cells)on Day 0 and 30, two times of blood sampling on day of 0 and 60 respectively for EV71 neutralizing antibody detection.The vaccine was manufactured by Institute of Medical Biology Chinese Academy of Medical Sciences.
  Interventions: Biological: EV71 inactived vaccine（Human diploid cells）
- Sequential vaccination group A (Experimental): One dose injection of EV71 inactived vaccines(Vero cells) on Day 0，following one dose of EV71 vaccine(EV71 inactived vaccines(human diploid cells), and two times of blood sampling on day of 0 and 60 respectively for EV71 neutralizing antibody detection.
  Interventions: Biological: EV71 inactived vaccine（Vero cells）; Biological: EV71 inactived vaccine（Human diploid cells）
- Sequential vaccination group B (Experimental): One dose injection of EV71 inactived vaccines(human diploid cells)on Day 0，following one does of EV71 vaccine(Sinovac Vaccine Technology Co., Ltd), and two times of blood sampling on day of 0 and 60 respectively for EV71 neutralizing antibody detection.
  Interventions: Biological: EV71 inactived vaccine（Vero cells）; Biological: EV71 inactived vaccine（Human diploid cells）

INTERVENTIONS:
Biological: EV71 inactived vaccine（Vero cells） — The EV71 inactived vaccine（Vero cells） was manufactured by Sinovac Biotech Co., Ltd.
  Arms: Sequential vaccination group A; Sequential vaccination group B; Single vaccine group A
Biological: EV71 inactived vaccine（Human diploid cells） — The EV71 inactived vaccine（Human diploid cells） was manufactured by Institute of Medical Biology Chinese Academy of Medical Sciences.
  Arms: Sequential vaccination group A; Sequential vaccination group B; Single vaccine group B

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of sequential vaccination of two EV71 inactived vaccines in healthy infants aged 6-35 months.

DETAILED DESCRIPTION:
This study is a opened,randomized and controlled phase Ⅳ clinical trial. The purpose of this study is to evaluate the immunogenicity and safety of sequential vaccination of two EV71 inactived vaccines in healthy infants aged 6-35 months. EV71 inactived vaccines(Vero cells）was manufactured by Sinovac Biotech Co., Ltd and EV71 inactived vaccines(Human diploid cells）was manufactured by Institute of Medical Biology Chinese Academy of Medical Sciences.300 infants aged between 6-35 months will be randomly assigned into experimental group in the ratio 1:1:1:1.The experimental group 1 received two doses EV71 inactived vaccines(Vero cells）on day 0 and 30. The experimental group 2 received two doses EV71 inactived vaccines (Human diploid cells）on day 0 and 30. The experimental group 3 received one dose EV71 inactived vaccines (Vero cells）on day 0 and one dose EV71 inactived vaccines (Human diploid cells）on day 30.The experimental group 4 received one dose EV71 inactived vaccines (Human diploid cells）on day 0 and one dose EV71 inactived vaccines (Vero cells）on day 30. To evaluate the immunogenicity of the vaccine, venous blood will be collected for the EV71 neutralizing antibody detection prior to vaccination and 30 days after the 2nd dose vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer aged 6-35 months;
* Proven legal identity;
* Guardians of the participants should be capable of understanding the written consent form, and such form should be signed before the infant being included into this study.

Exclusion Criteria:

* Prior vaccination with EV71 vaccine;
* History of hand，foot and mouth disease;
* Allergy to gentamicin; history of allergy to any vaccine or vaccine ingredient, or serious adverse reaction(s) to vaccination, such as urticaria,difficulty in breathing, angioneurotic edema, pain, etc;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc;
* Autoimmune diseases or immunodeficiency/immunosuppression;
* Severe neurological disorders (epilepsy, convulsions or convulsions) or psychosis;
* History of thyroidectomy, absence of spleen, functional absence of spleen, and any circumstances leading to absence of spleen or splenectomy;
* Diagnosed coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities) , or obvious bruising or coagulation disorders;
* Any immunosuppressant, cytotoxic medicine, or inhaled corticosteroids (except corticosteroid spray for treatment of allergic rhinitis or corticosteroid treatment on surface for acute non-complicated dermatitis) in the past 6 months;
* Receipt of any of the following products:

  1. Blood product within 3 months prior to study entry;
  2. Any live attenuated vaccine within 14 days prior to study entry;
  3. Any subunit vaccine or inactivated vaccine within 7 days prior to study entry;
  4. Any other study drugs within 30 days prior to study entry;
* Acute disease or acute stage of chronic disease within 7 days prior to study entry;
* Axillary temperature > 37.0℃;
* Any other factor that suggesting the volunteer is unsuitable for this study based on the opinions of investigators.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
The seroconversion rates (SCR) of the EV71 neutralizing antibody calculated based on the cutoff value of 1:8. | 30 days after two doses
  Subjects whose pre-immune EV71 antibody level < 1:8 and post-immune antibody level ≥ 1:8, or those whose pre-immune antibody level ≥ 1:8 and the increase of post-immune EV71 antibody level ≥ 4 folds are considered seroconverted

SECONDARY OUTCOMES:
The incidences of adverse reactions after each does | 0-30 days after each dose
  After each dose, a 30-minute safety observation will be conducted immediately. The body temperature, solicited local and general adverse events (AE) on day 0-7 were reported. Unsolicited adverse events on day 0-30 were also reported. Each AE case will be reviewed by the investigator to determine whether or not it was an adverse reaction (The vaccination-related AE).
The incidence of solicited local and general adverse events after each does | 0-7 days after each dose
  After each dose, a 30-minute safety observation will be conducted immediately. The body temperature, solicited local and general adverse events (AE) on day 0-7 were reported. Each AE case will be reviewed by the investigator to determine whether or not it was an adverse reaction (The vaccination-related AE).
Incidence of serious adverse events (SAEs) during the period of safety monitoring | 0-30 days after each dose
  Serious adverse events (SAEs) will be collected during the period of safety monitoring after each dose.
EV71 neutralizing antibody positive rate of each group after two doses. | 30 days after two doses
  Subjects whose post-immune antibody level ≥ 1:8 are considered antibody positive.
The Geometric mean titer (GMT) of the EV71 neutralizing antibody | 30 days after two doses
  The GMT 30 days of each group after two doses.
The geometric mean fold increase (GMI) of the EV71 neutralizing antibody | 30 days after two doses
  The GMI 30 days of each group after two doses.

CONTACTS AND LOCATIONS:
Overall Officials: AIqiang Xu, Principal Investigator — Shandong Provincal Center for Disease Control and Preventione
Locations (1):
- Rushan City Center for Disease Control and Prevention, Xiacun, Shandong, China

REFERENCES:
- [Derived] Xu Q, Cao Q, Yang W, Liu X, Liu H, Tian X, Li J, Fang X, Jia N, Zeng G, Xu A. Interchangeability of two Enterovirus 71 inactivated vaccines in Chinese children: A phase IV, open-label, and randomized controlled trial. Vaccine. 2020 Mar 10;38(12):2671-2677. doi: 10.1016/j.vaccine.2020.02.013. Epub 2020 Feb 14. PMID 32067817